CLINICAL TRIAL: NCT05122845
Title: Constitutive Study of a Serum Bank and Plasma Bank of Healthy Subjects Comparators to Dialysis Subjects (SPSSCD)
Acronym: SPSSCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: European Clinical Trial Experts Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018-A00040-55
Record Dates: First submitted 2021-10-19; First posted 2021-11-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Serum Bank; Plasma Bank; Dialysis
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy volunteers comparators to dialysis subjects (Experimental): Creation of a biological collection for biological analysis
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample — Blood test (10 tubes of 5mL) :
  - 6 tubes for : complete blood count, platelets, reticulocyte count, TP-INR, AST, ALT, GGT ferritin, serum iron, CRP, transferrin, soluble transferrin receptors, transferrin saturation coefficient enzymatic creatinine, MDRD, ionogram calcemia, phosphoremia, PTH, 25 (OH) D3, 1.25 (OH) 2D3.
  2 dry tubes 2 tube EDTA

SUMMARY:
To be able to evaluate the predictive value of glycosylated ferritin as a predictive marker of hepatic iron stock in dialysis patients, we need to validate these results with a cohort of healthy volunteers.

DETAILED DESCRIPTION:
This biological collection will include a sample of 2 dry tubes and 2 EDTA tubes. A haematological assessment (CBC, platelets, reticulocytes, Chr (hemoglobin content of reticulocytes), TP-INR, AST, ALT, GGT), measurement of biological markers of iron metabolism (ferritin, serum iron, CRP, transferrin, soluble receptors transferrin, transferrin saturation coefficient) as well as a creatinine assay to validate the normality of renal function in healthy volunteers (GFR established from the MDRD formula), a complete ionogram and a phosphocalcic balance being given the interactions in the dialysis patient (but also in normal subjects) between iron metabolism and phosphocalcic metabolism (calcemia, phosphoremia, PTH, 25OHD3, 1,25OH2D3) will be performed.

We will also study the links between iron overload in dialysis patients and the modulation of the synthesis of parathyroid hormone (intact PTH), FGF23, alpha Klotho and sclerostin.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age over 18 years old
* Healthy volunteers
* Having given their informed consent in writing
* Absence of current pathology
* No current treatment (except contraception)

Exclusion Criteria:

* Refusal of consent or absence of signature
* Minor, subject protected by law, (guardianship or curatorship, administrative protection measure)
* Pregnant woman, parturient
* Subject suffering from a condition liable to modify his blood parameters

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-23 (Actual)

PRIMARY OUTCOMES:
Number of participant with a serum and plasma bank creation | one day
  it is only a serum and plasma bank constitution

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Claude Galien, Quincy-sous-Sénart, France